CLINICAL TRIAL: NCT06122025
Title: Evaluating the Feasibility, Benefits and Acceptability to Patients and Health Care Professionals of Providing Secure Access of Linked Secondary Care and Patient's Personal Health Records in Cystic Fibrosis (CF)
Brief Title: Evaluation of Patient Access to People With Cystic Fibrosis (CF) and Healthcare Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Collaborators: University of Leeds (Other); Cystic Fibrosis Trust (Other); Leeds Beckett University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Patient Access V1.0, 12-JUN-17
Record Dates: First submitted 2023-10-20; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention [access to electronic healthcare records; EHR] (Active Comparator): For those in the intervention group, the participant will receive personalised access to their secondary electronic healthcare record (EHR) for 6 months. Individual access will be activated by the clinical team at the start of the study and will include views for;
  1. Current problems
  2. Current medication
  3. Test requests
  4. Letters
  5. Consultations
  6. Allergies
  7. Immunisations
  Interventions: Device: Patient Access
- Control [no access] (No Intervention): For those in the control group, participants will not receive access to their electronic healthcare record for the 6 month period. After the study, participants in the control group will have the opportunity to have access to their healthcare records

INTERVENTIONS:
Device: Patient Access — A 6-month pilot prospective interventional study with an independent groups design.
  Arms: Intervention [access to electronic healthcare records; EHR]

SUMMARY:
Cystic fibrosis (CF) is one of the most common inherited conditions in the United Kingdom (UK). There are 10,810 people living with CF in the UK, with median predicted survival now 47 years old. People with CF have multiple medical treatments to do on a daily basis, and the treatment burden is increasing. Adherence to treatment plays an important role in health outcomes and survival in CF.

Online access to their own health care records gives people an increased control over their own health, greater understanding of their conditions and has a potential to improve adherence to care plans and medications. Whilst implementation of electronic records is established in primary care, there has been a much poorer roll out of electronic care records in the secondary care system.

Leeds Teaching Hospitals CF Unit is a regional centre with around 650 adult and paediatric registered patients. Handwritten and typed paper records of patients under the care of the CF unit in Leeds were replaced in 2007 by electronic healthcare records (EHR; EMIS®). Patients view and obtain graphical feedback at each clinic visit including trends in parameters such as lung function, weight and inflammatory markers. In partnership with Egton Medical Information Systems (EMIS) web (EMIS®), a modification allowing secondary care access to patient records has been developed.

In a structured programme of research, the Leeds Adult CF Unit have firstly evaluated the implementation of the EHR in secondary care in terms of service delivery and cost improvement. In the second phase, the investigators sought patient feedback regarding which aspects of their EHR people with CF wish to access, and their priorities for development. This has informed the third phase in which the aim is to explore the impact of patient access to their EHR.

The aims of the trial are 1. To evaluate the feasibility, benefits and acceptability to patients and health care professionals of providing secure access of linked secondary care and patient's Personal Health Records in CF, and 2. To explore technological usability, future functionality and the impact of the shared records on clinical resources, communication and patient and health care professional satisfaction.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is one of the most common inherited conditions in the United Kingdom (UK). There are 10,810 people living with CF in the UK with median predicted survival now 47 years old. Patients with CF have multiple medical treatments to do on a daily basis, and the treatment burden is increasing. Adherence to treatment plays an important role in health outcomes and survival in CF.

Online access to their own health care records gives patients an increased control over their own health, greater understanding of their conditions and has a potential to improve adherence to care plans and medications. Other potential benefits include improved patient and multi-disciplinary team relationships, individual empowerment, satisfaction, time saving, transparency, shared decision making, positive behavioural change and opportunities for education.

The National Information Board launched an action framework in 2014 for personalised health and care 2020 by providing patients access to their electronic health records and work towards a patient centred healthcare in the UK and push towards a paperless National Health Service (NHS). But even today in 2017, paper still plays a major role throughout the NHS. Whilst implementation of electronic records is established in primary care, there has been a much poorer roll out of electronic care records in the secondary care system.

Leeds Teaching Hospitals CF Unit is a regional centre with around 650 adult and paediatric registered patients. Handwritten and typed paper records of patients under the care of the CF unit in Leeds were replaced in 2007 by electronic healthcare records (EHR; EMIS®). Patients view and obtain graphical feedback at each clinic visit including trends in parameters such as lung function, weight and inflammatory markers.

In partnership with Egton Medical Information Systems (EMIS) web (EMIS®), a modification allowing secondary care access to patient records has been developed. New Functionality in the Leeds CF EHR has the potential of delivering seamless data flow and feedback between patients and health care professionals. These new functionalities include full patient access to their personalised secondary care record as well as the ability to share a personalised patient generated record. Access to the secondary care record can be modified to include different views including current problems, current medication, test requests, letters, consultations, allergies and immunisations.

In a structured programme of research, the Leeds Adult CF Unit have firstly evaluated the implementation of the EHR in secondary care in terms of service delivery and cost improvement. In the second phase, the team sought patient feedback regarding which aspects of their EHR people with CF wish to access, and their priorities for development. This has informed the third phase in which the aim is to explore the impact of patient access to their EHR.

The aims of the trial are 1. To evaluate the feasibility, benefits and acceptability to patients and health care professionals of providing secure access of linked secondary care and patient's Personal Health Records in CF, and 2. To explore technological usability, future functionality and the impact of the shared records on clinical resources, communication and patient and health care professional satisfaction.

ELIGIBILITY:
Currently, there are approximately 400 people with cystic fibrosis (CF) attending the Regional Leeds Adult CF Unit, St James' University Hospital, Leeds, UK, and registered on the electronic healthcare record (EHR). Of these 400 patients, 100 people with CF will be recruited.

Inclusion criteria

* Diagnosis of CF (confirmed via genetic testing or sweat chloride tests)
* Aged 17 years and over
* Males and females
* Able to give written informed consent
* Records stored electronically on the EHR system at the Regional Leeds Adult CF Unit

Exclusion criteria

• Taking part in a clinical trial which prohibits patients taking part in other research

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
levels of anxiety | 6 months
  The effect on levels of anxiety of people with CF as measured by changes in the General Anxiety Disorder-7 (GAD-7) questionnaire.
  This questionnaire consists of 7 items (and one non-scored item which assigns weight to the degree to which anxiety problems have affected the patient's level of function), assessing over the last 2 weeks, how often patients have been bothered by anxiety related problems. Possible scores range from 0 (not at all) to 3 (nearly every day), with total scores of 0-5, 6-10. 11-15, and 15-21 representing mild, moderate, moderately severe and severe anxiety respectively.
levels of quality of life | 6 months
  The effect on quality of life of people with CF as measured by changes in the Cystic Fibrosis Questionnaire-Revised (CFQ-R) questionnaire.
  The CFQ-R is a disease-specific health-related qualify of life measure for people with CF and has undergone extensive reliability and validity testing. This questionnaire consists of 50 items, and assesses the following domains; Physical Functioning, Vitality, Health Perceptions, Respiratory Symptoms, Treatment Burden, Role Functioning, Emotional Functioning, and Social Functioning. Scores ranged from 0 to 100, with higher scores indicating better health-related qualify of life.

SECONDARY OUTCOMES:
levels of depression | 6 months
  The effect on levels of depression of people with CF as measured by changes in the Patient Health Questionnaire-9 (PHQ-9) questionnaire.
  The questionnaire is a brief (9 scored items and a non-scored item which assigns weight to the degree to which depressive problems have affected the patient's level of function) and multipurpose instrument for screening, diagnosing, measuring and monitoring the severity of depression in the past 2 weeks. Possible scores range from 0 (not at all) to 3 (nearly every day), with total scores of 0-5, 6-10. 11-15, and 15-21 representing mild, moderate, moderately severe and severe depression respectively.
Self-efficacy | 6 months
  Self-efficacy of people with CF as measured by changes in the Self-Efficacy to Manage Chronic Disease Scale (SEMCD) questionnaire.
  The 6 item scale covers several domains that are common across many chronic diseases; symptom control, role function, emotional functioning and communicating with physicians.
  The questionnaire asks participants how confident they are in doing certain activities. Responses are on a Likert scale from 1 (not very confident) to 10 (very confident). Participants choose a number that corresponds to their confidence that they can do the tasks regularly at the present time. The score for the scale is the mean of the six items; higher numbers reflect greater self efficacy.
Patient motivation towards health and care | 6 months
  Patient motivation towards health and care of people with CF as measured by changes in the Patient Activation Measure -13 (PAM-13) questionnaire.
  The questionnaire is a validated, commercially licenced tool (a US company, Insignia Health LLC) and consists of 13 items. Scores range between 0 and 100; the resulting score places the individual at one of four levels of activation:
  * Level 1 (0-25): Individuals tend to be passive and feel overwhelmed by managing their own health and may not understand their role in the care process
  * Level 2 (26-50): Individuals may lack the knowledge and confidence to manage their health
  * Level 3 (51-75): Individuals appear to be taking action but may still lack the confidence and skill to support their behaviours
  * Level 4 (76-100): Individuals have adopted many of the behaviours needed to support their health but may not be able to maintain them in the face of life stressors
Patient and provider relationships | 6 months
  Patient and provider relationships of people with CF as measured by changes in the Perceived Efficacy in Patient-Physician Interaction Questionnaire (PEPPI) questionnaire.
  The questionnaire consists of 10 items, and assesses the participants' level of trust in and interactions with their healthcare professionals (5 items on a scale of 0-5; not at all confident to very confident) and levels of self-efficacy (confidence) in self-care and self-management (5 items on a scale of 0-10; not at all confident to very confident). The total score is obtained by summing item scores, ranging from 10-50, with 50 representing high patient perceived self efficacy.
Computer literacy | 6 months
  Computer literacy of people with CF as measured by changes in an in-house questionnaire (questions taken from 'My Diabetes, My way' Questionnaire). It consists of 7 items related to computer literacy including the types, frequency, and experience of computer/internet use.
Perceptions of and intention to engage with patient access | 6 months
  Perceptions of and intention to engage with patient access by people with CF as measured by changes in an in-house questionnaire (derived from several previous questionnaires, some of which are theory driven).
  The questionnaire has 3 sections:
  * Section I has 9 items and asks questions about what people with CF think about having access to their electronic healthcare record and reasons for accessing, and not accessing, their record.
  * Section II has 11 items and asks questions about how might having access to their electronic healthcare record affect them. The responses in Section II are Likert, on a scale from Disagree to Agree, and also includes the option of 'Don't know'.
  * Section III has 18 items, based on the drivers and barriers to patients' acceptance of patient access, with responses of strongly disagree (1) to strongly agree (5).
System Usability Scale (SUS) | 6 months
  Patient access system usability as measured by changes in the System Usability Scale (SUS). It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree.
  The questionnaire consists of 10 items using Likert responses. Participants will rank each question from 0 to 4 based on how much they agree with each of the 10 statements; 4 means they agree completely, 0 means they disagree vehemently.
  For items 1, 3, 5, 7, and 9 the score contribution is the scale position minus 1. For items 2,4,6,8 and 10, the contribution is 5 minus the scale position. Scores for each question then added together and then multiplied by 2.5 to convert the original scores (0-40) to obtain the overall value of usability scale (0-100). Although the scores are 0-100, these are not percentages; a SUS score above a 68 would be considered above average and anything below 68 is below average.
Usability of the Patient Access system | 6 months
  Patient access system usability as measured by changes in the Perceived Health Web Site Usability Questionnaire (PHWSUQ)
  The PHWSUQ has 12 items on a 7-point Likert scale, and assesses three usability dimensions: satisfaction (very unsatisfied to very satisfied), ease of use (strongly disagree to strongly agree), and usefulness (strongly disagree to strongly agree). The questionnaire was modified to exclude two items relating to satisfaction as these are not relevant to patient access; ease of listening to audio-information, and quality of video information.
  Satisfaction scores range between 4 - 28, ease of use scores range between 3 - 21 and usefulness scores range between 3 - 21; higher scores reflect better usability.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Peckham, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

REFERENCES:
- [Derived] Chadwick HK, Sawant A, White H, Gillgrass L, Spoletini G, Clifton IJ, Etherington C, Peckham DG. Providing Mobile Patient Access to Their Electronic Secondary Care Patient Record in Adults With Cystic Fibrosis: Results of a Prospective, Parallel, Randomized Open-Pilot Quantitative Study. JMIR Form Res. 2025 Dec 25;9:e69747. doi: 10.2196/69747. PMID 41447265